CLINICAL TRIAL: NCT00130910
Title: Randomized, Double Blind, Placebo Controlled Trial of Albendazole in Soil-Transmitted Helminth and HIV-1 co-Infected Kenyan Individuals to Determine the Effect of Such Treatment on HIV-1 Disease Progression and Genital Shedding.
Brief Title: Treatment of Helminth co-Infection: Short-Term Effects on HIV-1 Progression Markers and Immune Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenya Medical Research Institute (Other); University of Nairobi (Other); Kenyatta National Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-1127-D03; NIH 5 P30 AI027757-19; UW Royalty Research Fund #3335
Record Dates: First submitted 2005-08-12; First posted 2005-08-16 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-11

CONDITIONS: HIV Infections; Helminthiasis
Keywords: HIV; Helminthiasis; Co-infection; Intestinal immune activation; Treatment Naive
MeSH Terms: conditions — HIV Infections; Helminthiasis; Coinfection | interventions — Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Albendazole
  Interventions: Drug: Albendazole
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albendazole — Albendazole 400mg x 3 first dose observed
  Other Names: Zentel
  Arms: 1
Drug: Placebo — Albendazole Placebo 400mg x 3 first dose observed
  Arms: 2

SUMMARY:
Identifying methods to slow disease progression in patients with HIV-1 infection remains a top priority in many regions of the world. In many countries, medications known to slow progression are not readily affordable or available. Many of the individuals living in these countries are also co-infected with a variety of other diseases such as tuberculosis, malaria and soil-transmitted helminths. There are data to suggest that infection with these agents may activate the immune system in HIV-1 co-infected individuals and may lead to more rapid HIV disease progression. This study will evaluate the potential impact of treating helminths in HIV-1 seropositive individuals. Markers of disease progression and immune activation will be assessed. We will also measure the amount of virus in genital secretions to determine if treatment of co-infection can reduce the infectiousness of HIV in these individuals.

DETAILED DESCRIPTION:
Many HIV infected individuals live in crowded urban settings. These conditions are associated with repeated intestinal parasite infections (helminths), which may alter the immune system in individuals with HIV and AIDS. This alteration in the immune system may increase both the susceptibility to other infections and the severity of these infections in these individuals. Prior studies have shown that in HIV infected individuals, intestinal parasites are associated with increased levels of the HIV virus circulating in the blood. Studies have also clearly shown that in individuals with HIV, progression to AIDS can be predicted by the quantity of HIV virus detectable within the blood. It is important to determine whether treating helminth co-infection in patients with HIV will help individuals control HIV infection and slow disease progression.

The investigators propose a study to characterize the short-term effect of antihelminth therapy on HIV disease progression, markers of immune activation and levels of HIV in genital secretions. They also plan to determine the prevalence of helminth infection in individuals with HIV. This study will examine factors that might affect an individual's risk of helminth infection, such as CD4 count, viral load, age, gender and duration of time spent in an urban setting. In addition, the investigators will conduct a randomized clinical trial to determine the effect of treating helminth infection on markers of immune activation, HIV disease progression and risk of transmission as measured by HIV-1 RNA in genital secretions. The study will be conducted in a group of HIV infected individuals in and around Nairobi, Kenya who do not yet meet criteria for highly active antiretroviral therapy (HAART).

Identifying inexpensive and practical methods to delay HIV progression offers tremendous public health benefits. At the present time, highly active antiretroviral therapy is being rapidly scaled up in resource poor settings. The demand for these drugs currently far outweighs the capacity for such services to be provided in many regions. For the millions of people infected by HIV in resource poor settings, delaying immunosuppression for months to years could allow important developments in infrastructure which would permit the maximum number of individuals to benefit from highly active antiretroviral therapy.

HIV-1 infected adults will be invited to participate in the trial. Women whose pregnancy test is positive will be excluded from the study. A physical examination will be conducted on all prospective clients, and those found to have clinical pallor, or signs and symptoms of active tuberculosis, malaria or malignancy will be excluded from the study. Individuals with CD4 counts greater than 250 cells/mm3 will be enrolled in the study following written informed consent.

HIV-1 infected patients who meet inclusion and exclusion criteria will be enrolled for screening. Stool samples will be collected at enrollment and evaluated for ova and parasites. All patients who are found to have positive stool parasite examinations and who consent to participate will be enrolled in the treatment phase of the study. Those who are found to have negative stool specimens will not continue to the treatment phase. Baseline demographic and socio-economic data will be collected from these patients in order to evaluate the prevalence and correlates of helminth infection among HIV-1 infected individuals. Those who are found to be infected with helminths but who decline to participate in the treatment phase will be treated at no charge with a three day course of albendazole (400 mg/day) by the study investigators. Those patients who are enrolled in the treatment phase will have blood collected for baseline plasma HIV-1 RNA levels. Computer-generated random number allocation will be used to assign treatment group. The pharmacy at the Kenya Medical Research Institute will be responsible for the determination of randomization group and distribution of albendazole and placebo. The pharmacy will also be responsible for maintaining records regarding treatment group. Treatment will be provided in the form of a six 200 mg pills of albendazole or six placebo pills identical in appearance. Both placebo and albendazole will be provided in an identical appearing envelope. Treatment arms consist of either initial therapy with albendazole (400 mg per day for three days) or two placebo pills per day initially. All patients will be required to visit the clinic twelve weeks after enrollment. At this twelve week visit, stool samples will again be collected for evaluation of helminth infection. Plasma CD4 count and HIV-1 RNA level measurements will be repeated at this twelve week visit. All patients who received placebo initially as well as all patients with evidence of helminth infection will be treated with open-label albendazole therapy regardless of initial treatment arm. At enrollment and the twelve week visit, lymphocytes will also be isolated from serum samples for assessment of immune activation markers. Genital HIV-1 RNA levels will be compared in 100 individuals randomized to immediate versus deferred antihelminthics at baseline and at the 3-month visit (prior to receiving deferred therapy). This will provide data quantifying the potential effect of anti-helminthic treatment on genital HIV-1 RNA. Consenting adults will have genital swabs collected (semen or cervical/vaginal) and placed in freezing media prior to cryopreservation and transport to Fred Hutchinson Cancer Research Center for HIV-1 RNA assays.

Patients who do not follow-up as directed will be contacted by the administrative support team at their homes in order to determine the reason for each loss to follow up. Any adverse events during the treatment period will be reported and managed accordingly at the treatment clinic.

ELIGIBILITY:
Inclusion Criteria:

* Participants must not be or have been on highly active antiretroviral therapy.
* Participants must have a CD4 count greater than 250 cells/mm3.
* Participants must be at least 18 years of age.
* Participants must be able and willing to participate and give written informed consent.
* Participants must be able and willing to return for the scheduled follow-up visits.
* In addition, in order to be included in the treatment phase of the study, patients must have at least one stool specimen positive for a soil transmitted helminth.

Exclusion Criteria:

* Participants who have received treatment for helminth infection in the past 6 months (by self report or chart review).
* Participants must not be pregnant at the time of treatment (by urine HCG testing).
* Participants who present with other serious co-morbidities such as severe anaemia, malaria or tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2006-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change in markers of HIV-1 disease progression | 12 weeks
CD4 count | 12 weeks
HIV-1 RNA level | 12 weeks
Genital HIV-1 RNA levels | 12 weeks

SECONDARY OUTCOMES:
Immune activation markers of global T cell activation | 12 weeks
Numbers of CD4+ and CD8+ T cells expressing Ki67 | 12 weeks
Naïve and memory T cell subsets | 12 weeks
Type and number of helminth co-infections | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Judd L Walson, MD, MPH, Study Director — University of Washington; Grace C. John-Stewart, MD, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya

REFERENCES:
- [Background] 2004 report on the global AIDS epidemic : 4th global report. UNAIDS
- [Background] Fincham JE, Markus MB, Adams VJ. Could control of soil-transmitted helminthic infection influence the HIV/AIDS pandemic. Acta Trop. 2003 May;86(2-3):315-33. doi: 10.1016/s0001-706x(03)00063-9. PMID 12745148
- [Background] Elliott AM, Mawa PA, Joseph S, Namujju PB, Kizza M, Nakiyingi JS, Watera C, Dunne DW, Whitworth JA. Associations between helminth infection and CD4+ T cell count, viral load and cytokine responses in HIV-1-infected Ugandan adults. Trans R Soc Trop Med Hyg. 2003 Jan-Feb;97(1):103-8. doi: 10.1016/s0035-9203(03)90040-x. PMID 12886815
- [Background] Bentwich Z, Weisman Z, Moroz C, Bar-Yehuda S, Kalinkovich A. Immune dysregulation in Ethiopian immigrants in Israel: relevance to helminth infections? Clin Exp Immunol. 1996 Feb;103(2):239-43. doi: 10.1046/j.1365-2249.1996.d01-612.x. PMID 8565306
- [Background] Kassu A, Tsegaye A, Wolday D, Petros B, Aklilu M, Sanders EJ, Fontanet AL, Van Baarle D, Hamann D, De Wit TF. Role of incidental and/or cured intestinal parasitic infections on profile of CD4+ and CD8+ T cell subsets and activation status in HIV-1 infected and uninfected adult Ethiopians. Clin Exp Immunol. 2003 Apr;132(1):113-9. doi: 10.1046/j.1365-2249.2003.02106.x. PMID 12653845
- [Background] Elliott AM, Kyosiimire J, Quigley MA, Nakiyingi J, Watera C, Brown M, Joseph S, French N, Gilks CF, Whitworth JA. Eosinophilia and progression to active tuberculosis in HIV-1-infected Ugandans. Trans R Soc Trop Med Hyg. 2003 Jul-Aug;97(4):477-80. doi: 10.1016/s0035-9203(03)90096-4. PMID 15259486
- [Background] Olsen A. The proportion of helminth infections in a community in western Kenya which would be treated by mass chemotherapy of schoolchildren. Trans R Soc Trop Med Hyg. 1998 Mar-Apr;92(2):144-8. doi: 10.1016/s0035-9203(98)90721-0. PMID 9764316
- [Background] Wolday D, Mayaan S, Mariam ZG, Berhe N, Seboxa T, Britton S, Galai N, Landay A, Bentwich Z. Treatment of intestinal worms is associated with decreased HIV plasma viral load. J Acquir Immune Defic Syndr. 2002 Sep 1;31(1):56-62. doi: 10.1097/00126334-200209010-00008. PMID 12352151
- [Background] Lawn SD, Karanja DM, Mwinzia P, Andove J, Colley DG, Folks TM, Secor WE. The effect of treatment of schistosomiasis on blood plasma HIV-1 RNA concentration in coinfected individuals. AIDS. 2000 Nov 10;14(16):2437-43. doi: 10.1097/00002030-200011100-00004. PMID 11101053
- [Background] Bennett A, Guyatt H. Reducing intestinal nematode infection: efficacy of albendazole and mebendazole. Parasitol Today. 2000 Feb;16(2):71-4. doi: 10.1016/s0169-4758(99)01544-6. PMID 10652492
- [Derived] Walson JL, Stewart BT, Sangare L, Mbogo LW, Otieno PA, Piper BK, Richardson BA, John-Stewart G. Prevalence and correlates of helminth co-infection in Kenyan HIV-1 infected adults. PLoS Negl Trop Dis. 2010 Mar 30;4(3):e644. doi: 10.1371/journal.pntd.0000644. PMID 20361031
- [Derived] Walson JL, Otieno PA, Mbuchi M, Richardson BA, Lohman-Payne B, Macharia SW, Overbaugh J, Berkley J, Sanders EJ, Chung MH, John-Stewart GC. Albendazole treatment of HIV-1 and helminth co-infection: a randomized, double-blind, placebo-controlled trial. AIDS. 2008 Aug 20;22(13):1601-9. doi: 10.1097/QAD.0b013e32830a502e. PMID 18670219